CLINICAL TRIAL: NCT06163040
Title: Empliciti® (Elotuzumab) Post-Marketing Surveillance Study for Patients With Multiple Myeloma in Taiwan
Brief Title: A Study to Evaluate the Safety of Empliciti® (Elotuzumab) When Treating Patients With Multiple Myeloma in Taiwan
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA204-219
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Relapsed or Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — elotuzumab; pomalidomide; Dexamethasone; Lenalidomide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treated with Elotuzumab in combination with pomalidomide and dexamethasone
  Interventions: Drug: Elotuzumab in combination with pomalidomide and dexamethasone
- Treated with Elotuzumab in combination with lenalidomide and dexamethasone
  Interventions: Drug: Elotuzumab in combination with lenalidomide and dexamethasone

INTERVENTIONS:
Drug: Elotuzumab in combination with pomalidomide and dexamethasone — Participants who received elotuzumab in combination with pomalidomide and dexamethasone for RRMM and had ≥2 prior lines of therapy (including lenalidomide and a proteasome inhibitor)
  Groups: Treated with Elotuzumab in combination with pomalidomide and dexamethasone
Drug: Elotuzumab in combination with lenalidomide and dexamethasone — Participants who received elotuzumab in combination with pomalidomide and dexamethasone for RRMM and had ≥2 prior lines of therapy (including lenalidomide and a proteasome inhibitor)
  Groups: Treated with Elotuzumab in combination with lenalidomide and dexamethasone

SUMMARY:
This observational study aimed to assess the safety of elotuzumab when used in combination with pomalidomide and dexamethasone for the treatment of relapsed and refractory multiple myeloma (RRMM) in participants who had received at least two prior therapies, including lenalidomide and a proteasome inhibitor. The study will also assess the safety of elotuzumab when used in combination with lenalidomide and dexamethasone in RRMM participants who had received one to three prior therapies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Confirmed diagnosis of RRMM
* Received ≥ 2 prior therapies including lenalidomide and a proteasome inhibitor
* Planning to receive elotuzumab in combination with pomalidomide and dexamethasone at physician's medical judgement OR
* Age ≥ 18 years
* Confirmed diagnosis of RRMM
* Received one to three prior therapies
* Planning to receive elotuzumab in combination with lenalidomide and dexamethasone at physician's medical judgement

Exclusion Criteria:

* Participants with therapeutic indications for which elotuzumab in combination with pomalidomide/lenalidomide and dexamethasone has not been approved in Taiwan
* Participants who are contraindicated for treated with elotuzumab in combination with pomalidomide/lenalidomide and dexamethasone (as described in the Taiwan label)
* Participants who participate in other interventional clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (≥ 18 years of age) patients who have a confirmed diagnosis of RRMM, who 1) have received at least 2 prior therapies, including lenalidomide and a proteasome inhibitor, and are planning to receive Empliciti in combination with pomalidomide and dexamethasone, or 2) have received one to three prior therapies and are planning to receive Empliciti in combination with lenalidomide and dexamethasone
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2023-12-22 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2025-03-17 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | 25 weeks from start of treatment, or during a 30-day follow-up period following treatment discontinuation (whichever time period falls at a later date)
  Assessed according to NCI CTCAE v5.0
Number of participants with adverse events of special interest | 25 weeks from start of treatment, or during a 30-day follow-up period following treatment discontinuation (whichever time period falls at a later date)
  Opportunistic infections including viral hepatitis and tuberculosis reactivation

SECONDARY OUTCOMES:
Number of participants with fungal infections | 25 weeks from start of treatment, or during a 30-day follow-up period following treatment discontinuation (whichever time period falls at a later date)
Number of participants with reactivation of viral hepatitis | 25 weeks from start of treatment, or during a 30-day follow-up period following treatment discontinuation (whichever time period falls at a later date)
Number of participants with other viral infection/reactivation | 25 weeks from start of treatment, or during a 30-day follow-up period following treatment discontinuation (whichever time period falls at a later date)
Number of participants with tuberculosis infection/reactivation | 25 weeks from start of treatment, or during a 30-day follow-up period following treatment discontinuation (whichever time period falls at a later date)
Number of participants with other opportunistic infections | 25 weeks from start of treatment, or during a 30-day follow-up period following treatment discontinuation (whichever time period falls at a later date)
Number of participants with lymphopenia | 25 weeks from start of treatment, or during a 30-day follow-up period following treatment discontinuation (whichever time period falls at a later date)
  Laboratory abnormality and/or adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- Taiwan (4):
  - Chang Gung Memorial Hospital- Chiayi, Chiayi City, Chiayi
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
  - China Medical University Hospital, Taoyuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts